CLINICAL TRIAL: NCT05150288
Title: Growth and Feeding Tolerance of Infants Consuming a Formula Supplemented With Human Milk Oligosaccharides (HMOs): An Uncontrolled, Open-label, Prospective Study
Brief Title: Human Milk Oligosaccharides (HMOs) Post-market Study on Infants (NEHMO)
Acronym: NeHMO DACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Waldkrankenhaus Protestant Hospital, Spandau (Other); Kinderarztpraxis Köllges, Mossakowski und Meyer-Krott, Mönchengladbach (Unknown); Gemeinschaftspraxis Kinder- und Jugendpraxis Dr. Stepan Dreher und Tina Hübler, Geldern (Unknown); Kinder- und Jugendarzt Dr. Umpfenbach und Dr. Lorenz, Viersen (Unknown); Kinder- und Jugendärztliche Gemeinschaftspraxis Bedikian & Bouikidis, Oberhausen (Unknown); Kinderarztpraxis Dr. Zakarian, Düsseldorf (Unknown); Facharztpraxis für Kinder- und Jugendmedizin Dr. Aulinger, Burglengenfeld (Unknown); Zentrum für Kinder- und Jugendgesundheit Regensburg (Unknown); Kinder- und Jugendarztpraxis Schwabach (Unknown); Praxis Dr. Klee, Bürstadt (Unknown); Facharzt für Säuglings-, Kinder- und Jugendmedizin, Bremen (Unknown); Praxis Al-Radhi, Ehingen (Unknown); Kinder und Jugendarztpraxis Dr. Maier, Leinfelden-Echterdingen (Unknown); Kinder- und Jugendarztpraxis Dr. Kröckel, Dr. Ciesla, Berlin (Unknown); Facharzt für Kinder- und Jugendheilkunde Dr. Faustmann, Oberwart (Unknown); Nestlé Research, Société des Produits Nestlé S.A., Lausanne, Switzerland (Unknown); Global Medical Affairs, Société des Produits Nestlé S.A., Vevey, Switzerland (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1806INF- DACH
Record Dates: First submitted 2021-11-25; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Growth; Tolerance; Adverse Event; Disorder of Intestine; Formula Satisfaction
Keywords: Growth; Tolerance; Adverse Event; Gastrointestinal tolerance; Infant formula; Human milk oligosaccharides; 2'-fucosyllactose; Lacto-N-neotetraose; Real-world
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Formula-fed infants (Experimental): Infants fed exclusively with experimental formula
  Interventions: Other: HMO-supplemented infant formula
- Mixed-fed infants (Experimental): Infants receiving breastmilk and experimental formula
  Interventions: Other: HMO-supplemented infant formula
- Breast-fed infants (No Intervention): Reference group of exclusively breastfed

INTERVENTIONS:
Other: HMO-supplemented infant formula — Starter Infant Formula supplemented with 1.5g/L of Human Milk Oligosaccharides
  Arms: Formula-fed infants; Mixed-fed infants

SUMMARY:
Human milk oligosaccharides (HMOs) represent the third largest solid component of breast milk. Technology advancements made it possible to supplement infant formulas with HMOs (2'FL, LNnT). Two published RCTs have demonstrated that infant formulas supplemented with 2'FL or 2'FL+LNnT are safe, well-tolerated, support normal grow, and may support healthy GI function and confer immune benefits. The performance of HMOs-supplemented formulas assessed in a real-world setting is complementary to previously conducted RCTs conducted in highly controlled clinical settings. Main objectives will be to monitor the safety & tolerance of HMOs-supplemented formulas in larger and diverse infant populations; to assess the performance of HMOs-supplemented formulas in mixed-fed infants, a population that was not studied in previous RCTs but likely represents a relatively common feeding regimen. Finally, considering the potential health/immune benefits of HMOs, it is also important explore the incidences of illnesses (i.e., respiratory illnesses, GI illnesses, and fever) associated with consuming HMOs-supplemented formulas and compare with breastfed infants data.

DETAILED DESCRIPTION:
Objectives:

The main objective of this study is to document the growth and feeding tolerance of healthy term infants consuming an infant formula supplemented with HMOs for 8 weeks (56 days), in a real-world setting.

Main endpoints:

1. Growth documented via monitoring the anthropometric parameters including weight, length, head circumference, BMI and their corresponding z-scores (i.e., z-scores for weight-for-age, length-for-age, weight-for-length, head circumference-for-age, and BMI-for-age) calculated using the 2006 WHO Growth Standards
2. Feeding tolerance assessed via monitoring parent-reported overall GI symptom burden measured by the Infant Gastrointestinal Symptom Questionnaire (IGSQ) index score (13-item summary score)

Additional objectives:

To describe the following outcomes in infants fed an infant formula supplemented with HMOs:

1. Formula acceptability
2. Despite there are no expected safety concerns, standard Adverse Events (AEs) monitoring will be implemented during the study

Additional endpoints:

1. Formula acceptability assessed by the Study Formula Satisfaction Questionnaire
2. Reported AEs and Serious Adverse Events (SAEs) including type, incidence, severity, seriousness and relation to study formula consumption as well as concomitant medications and non-pharmacological treatments.

   * Select morbidities of interest (i.e., respiratory illnesses, GI illnesses, and fever) will be collected as part of AE reporting and specific corresponding AE guidance forms will be used to standardize reporting of such AEs

Trial design:

Uncontrolled, single arm, open-label, prospective study in infants (enrolled at postnatal age 7 days to 2 months) fed the study formula for 8 weeks (56 days)

A group of exclusively breastfed infants (BF) will serve as a reference group in parallel to the study arm. For the BF group, Infants must have been exclusively consuming breast milk since birth, and their parent(s) must have made the decision to continue exclusively breastfeeding until at least 4 month of age

Trial population:

Healthy, male and female, term infants, 7 days postnatal age to 2 months of age at the enrollment

Treatment duration:

Total study participation/intervention up to approximately 8 weeks

ELIGIBILITY:
Inclusion Criteria:

* Evidence of personally signed and dated informed consent document indicating that the infant's parent(s) have been informed of all pertinent aspects of the study
* Parent(s) are willing and able to fulfill the requirements of the study protocol
* Healthy full term (37-42 weeks gestation) infant
* Be between post-natal age (Date of Birth = Day 0) 7 days to 2 months
* Parent(s) must have independently elected, before enrollment, to formula feed

Exclusion Criteria:

* Any known intolerance/allergy to cow's milk (formula-fed group only)
* systemic disorders (cardiac, respiratory, endocrinological, hematologic, gastointestinal, or other)
* conditions requireing infant feedings other than those specified in the protocol
* Infants must have been exclusively consuming breast milk since birth, and their parent(s) must have made the decision to continue exclusively breastfeeding until at least 4 month of age

Ages: 7 Days to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-07-24 (Actual)

PRIMARY OUTCOMES:
World Health Organization (WHO) based weight-for-age z-scores | 8 weeks (study end)
  Weight-for-age z-scores using WHO growth standards
World Health Organization (WHO) based length-for-age z-scores | 8 weeks (study end)
  Length-for-age z-scores using WHO growth standards
World Health Organization (WHO) head-circumference-for-age z-scores | 8 weeks (study end)
  head-circumference-for-age z-scores using WHO growth standards
World Health Organization (WHO) based body-mass-index (BMI)-for-age z-scores | 8 weeks (study end)
  Weight and height will be combined to calculate BMI in kg/m^2, then BMI-for-age z-scores will be derived using WHO growth standards
Feeding tolerance | 4 weeks (study midpoint)
  The Infant Gastrointestinal Symptom Questionnaire (IGSQ) index score will be used to assess GI distress. This is a validated 13-item questionnaire where each item is scored on a scale of 1 to 5 with higher values indicating greater GI distress. A composite IGSQ score is derived from summing the individual scores with a possible range of 13 to 65 where higher values indicate greater GI distress and values ≤23 indicate no digestive distress
Feeding tolerance | 8 weeks (study end)
  The Infant Gastrointestinal Symptom Questionnaire (IGSQ) index score will be used to assess GI distress. This is a validated 13-item questionnaire where each item is scored on a scale of 1 to 5 with higher values indicating greater GI distress. A composite IGSQ score is derived from summing the individual scores with a possible range of 13 to 65 where higher values indicate greater GI distress and values ≤23 indicate no digestive distress

SECONDARY OUTCOMES:
Formula acceptability | 4 weeks (study midpoint), 8 weeks (study end)
  Study Formula Satisfaction Questionnaire
Standard adverse events (AEs) reporting for safety assessment | From the time the informed consent form has been signed at enrollment infant age less than 7 days to 2 months through the 8 weeks of intervention
  Reported adverse events (AEs) and Serious Adverse Events (SAEs) include type, incidence, severity, seriousness and relation to feeding
Weight | 8 weeks (study end)
  Weight measurements in grams
Length | 8 weeks (study end)
  Length measurements in centimeters
Head circumference | 8 weeks (study end)
  Head circumference measurements in centimeters
Body-mass-index (BMI) | 8 weeks (study end)
  Weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Locations (17):
- Facharzt für Kinder- und Jugendheilkunde, Oberwart, Austria
- Germany (14):
  - Kinder- und Jugensarztpraxis, Berlin
  - Evangelisches Waldkrankenhaus Spandau, Berlin-Spandau
  - Facharzt für Säuglings-, Kinder- und Jugendmedizin, Bremen
  - Facharztpraxis für Kinder- und Jugendmedizin, Burglengenfeld
  - Praxis Dr. Klee, Bürstadt
  - Kinderarztpraxis, Düsseldorf
  - Praxis Al-Radhi, Ehingen
  - Gemeinschaftspraxis Kinder- und Jugendarztpraxis, Guelders
  - Kinder und Jugendarztpraxis, Leinfelden-Echterdingen
  - Kinderarztpraxis Köllges, Mönchengladbach
  - Kinder- und Jugendärztliche Gemeinschaftspraxis, Oberhausen
  - Zentrum für Kinder- und Jugendgesundheit, Regensburg
  - Kinder- und Jugendarztpraxis, Schwabach
  - Kinder- und Jugendarzt, Viersen
- Switzerland (2):
  - Nestlé Research, Société des Produits Nestlé S.A., Lausanne
  - Global Medical Affairs, Société des Produits Nestlé, Vevey

REFERENCES:
- [Background] Storm HM, Shepard J, Czerkies LM, Kineman B, Cohen SS, Reichert H, Carvalho R. 2'-Fucosyllactose Is Well Tolerated in a 100% Whey, Partially Hydrolyzed Infant Formula With Bifidobacterium lactis: A Randomized Controlled Trial. Glob Pediatr Health. 2019 Mar 15;6:2333794X19833995. doi: 10.1177/2333794X19833995. eCollection 2019. PMID 30906817